CLINICAL TRIAL: NCT03387176
Title: Efficacy of a Gluten-free Diet in Difficult to Manage Nephrotic Syndrome: Utility of Plasma Zonulin Levels as a Predictive Biomarker
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 17-01307
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- zonulin ≤17.5 ng/ml: Pediatric patients with difficult-to-manage nephrotic syndrome will be stratified based on the plasma zonulin concentration into two groups
  Interventions: Other: Implementation of a gluten-free diet
- zonulin >17.5 ng/ml: Pediatric patients with difficult-to-manage nephrotic syndrome will be stratified based on the plasma zonulin concentration into two groups
  Interventions: Other: Implementation of a gluten-free diet

INTERVENTIONS:
Other: Implementation of a gluten-free diet — Patients will be placed on gluten free diet for 9-12 months.

SUMMARY:
Elevated plasma zonulin levels, which are supportive of a diagnosis of CD (celiac disease) in children with gastrointestinal symptoms, may indicate patients with difficult-to-manage NS who will benefit from initiation of a GFD (gluten free diet). This pilot study will determine whether high plasma zonulin levels can be used as a screening tool to identify patients with NS (nephrotic syndrome) who are likely to demonstrate a beneficial response to a GFD. It will provide important information about the feasibility of testing the efficacy of a GFD for this condition and assist in the design and sample size calculation for a definitive trial to test the beneficial effect of this dietary intervention. Although NS is a rare condition in childhood, it is a chronic disease that can lead to short- and long-term disability especially in those with difficult-to-manage disease. There is an urgent need to develop safe and effective new therapies in this subgroup. This project may indicate the utility of a common dietary modification, a GFD, to treat these patients. The growing medical use of and greater access to gluten-free food items underscore the feasibility and timeliness of this approach.

ELIGIBILITY:
Inclusion Criteria:

* Steroid sensitive NS: complete remission of proteinuria in response to administration of a standard course of corticosteroids
* Difficult-to-manage NS: disease that cannot be controlled without incurring intolerable side effects from currently available immunosuppressive agents, namely corticosteroids, calcineurin inhibitors, mycophenolate mofetil, or rituximab. Patients with biopsy-proven MCD or FSGS will be eligible as long as they have steroid sensitive disease. However, a renal biopsy will not be required for enrollment into the trial.

Exclusion Criteria:

* Any patient diagnosed with nephrotic syndrome that is not considered steroid sensitive or frequently relapsing
* Pre-existing celiac disease or gastro-intestinal disorder that precludes use of a GFD

Ages: 9 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children age 9 months to 18 years of age with steroid sensitive Nephrotic Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Change in disease activity measured by relapse rate | 12 Months
  Response is defined as a ≥50%decrease in relapse rate
Change in disease activity measured by change in dosage of corticosteroids and immunosuppressive medications | 12 Months
  reduction by ≥1 drug in exposure to immunosuppressive medications in response to the GFD

CONTACTS AND LOCATIONS:
Overall Officials: Howard Trachtman, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States